CLINICAL TRIAL: NCT00166894
Title: Evaluation of the Triggering Receptor Expressed on Myeloid Cells-1 (TREM-1) as a Diagnostic Tool for Patients With Pleural Effusion
Brief Title: Use of the Triggering Receptor Expressed on Myeloid Cells-1 (TREM-1) in the Diagnosis of Pleural Effusion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700516
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-11-24 (Estimated); Status verified 2005-05

CONDITIONS: Pleural Effusion
Keywords: pleural effusion; TREM-1
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other

SUMMARY:
The aim of this trial is to evaluate the level of TREM-1 in different kinds of pleural effusion.

DETAILED DESCRIPTION:
The triggering receptor expressed on myeloid cells-1 (TREM-1) is a member of the immunoglobulin superfamily, and its expression is upregulated on phagocytic cells in the presence of bacteria or fungi. Several experiments by Bouchon and colleagues showed that TREM-1 mediates the acute inflammatory response to microbial products. Human tissues infected with bacteria are infiltrated with neutrophils and macrophages that express high levels of TREM-1. Conversely, TREM-1 is only weakly expressed in samples from patients with noninfectious inflammatory disorders. In addition, TREM-1 is shed from the membrane of activated phagocytes and can be found in a soluble form in body fluids. The presence of a soluble form of TREM-1 in samples of bronchoalveolar lavage fluid from mechanically ventilated patients has been shown to be a good indicator of infectious pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of pleural effusion
* Pleural effusion proved by chest sonography

Exclusion Criteria:

* Conditions for which thoracentesis are contraindicated
* Pregnancy

Min Age: 18 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Pan-Chyr Yang, MD, PhD, Principal Investigator — Department of International Medicine, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan